CLINICAL TRIAL: NCT05439707
Title: Effects of Perioperative Transauricular Vagus Nerve Electrical Stimulation on Postoperative Delirium, Postoperative Cognitive Dysfunction and Chronic Postsurgical Pain in Patients Undergoing Arthroplasty.
Brief Title: Effects of Perioperative Transauricular Vagus Nerve Electrical Stimulation on POD, POCD and CPSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Central Hospital (Other)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other); The First People's Hospital of Xuzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: XuzhouCH20220620
Record Dates: First submitted 2022-06-20; First posted 2022-06-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Delirium; Chronic Post Operative Pain
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The transaricular vagus nerve stimulator was placed in the left ear trunk, which is dominated only by the auricular branch of the vagus nerve. Continuous stimulation was performed at a frequency of 25Hz with pulse width of 300 μs. The stimulation was adjusted to be higher than the perception threshold and lower than the pain threshold. Each stimulation lasted for 30 minutes, three times per day (morning, noon, evening), from 1 day before surgery to 7 days after surgery, and the treatment lasted for 9 consecutive days.
  Interventions: Device: transaricular vagus nerve stimulation
- Control group (Sham Comparator): The transaricular vagus nerve stimulator was placed in the same position as the experimental group, covered with an insulating film and placed at the site of the stimulation, so that the patient could not actually receive the electrical stimulation. Continuous stimulation was performed at a frequency of 25Hz and pulse width of 300 μs, and the stimulation was adjusted to be higher than the perception threshold and lower than the pain threshold. Each stimulation lasted for 30 minutes, three times per day (morning, noon, evening), from 1 day before surgery to 7 days after surgery, for 9 consecutive days.
  Interventions: Device: fake transaricular vagus nerve stimulation

INTERVENTIONS:
Device: transaricular vagus nerve stimulation — The transaricular vagus nerve stimulator was placed in the left ear trunk, which is dominated only by the auricular branch of the vagus nerve. Continuous stimulation was performed at a frequency of 25Hz with pulse width of 300 μs. The stimulation was adjusted to be higher than the perception threshold and lower than the pain threshold. Each stimulation lasted for 30 minutes, three times per day (morning, noon, evening), from 1 day before surgery to 7 days after surgery, and the treatment lasted for 9 consecutive days.
  Arms: Experimental group
Device: fake transaricular vagus nerve stimulation — The transaricular vagus nerve stimulator was placed in the same position as the experimental group, covered with an insulating film and placed at the site of the stimulation, so that the patient could not actually receive the electrical stimulation. Continuous stimulation was performed at a frequency of 25Hz and pulse width of 300 μs, and the stimulation was adjusted to be higher than the perception threshold and lower than the pain threshold. Each stimulation lasted for 30 minutes, three times per day (morning, noon, evening), from 1 day before surgery to 7 days after surgery, for 9 consecutive days.
  Arms: Control group

SUMMARY:
Postoperative delirium (POD) and postoperative cognitive dysfunction (POCD) occur in 11-51% of patients after surgery, and its prevalence increases with age. The occurrence of delirium is associated with increased morbidity and mortality, prolonged hospital stay, worse functional recovery. Orthopedic procedures and specifically joint replacements have been considered as a major risk for development of chronic postsurgical pain (CPSP). Approximately 13-44% of patients will develop CPSP after knee or hip arthOpioid abuseroplasty. CPSP may cause the discomfort, distress, disability and opioid abuse. Mounting evidence has revealed that inflammation triggered by surgical trauma plays a key role in POD, POCD and CPSP. Recent studies found that vagus nerve stimulation showed the suppression of inflammation. In this study, the effect of perioperative transauricular vagus nerve stimulation on the prognosis of patients undergoing arthroplasty will be investigated, providing potential solutions for the prevention and treatment of postoperative cognitive dysfunction, postoperative delirium and chronic postsurgical pain.

DETAILED DESCRIPTION:
The investigators assessed POD by the Confusion Assessment Method for the ICU twice daily for 7 days after surgery. Participants' cognitive function was assessed with neuropsychological battery tests. The tests included digit span (forward and backward), Corsi block, paired associate verbal learning, digit symbol test, trail-making test and so on.The investigators make a CPSP diagnosis based on the 11th revision of the International Classification of Diseases.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 80 years old.
* ASA grade I-Ⅲ.
* elective knee or hip replacement.

Exclusion Criteria:

* Mini-Mental State Examination (MMSE) score < 23.
* Education years<7.
* Peptic ulcer disease, serious cardiac-cerebral vascular disease.
* Neurological or psychiatric disorders.
* History of drug and alcohol abuse.
* Hepatic and/or kidney dysfunction.
* BMI>35.
* Patients on antidepressants.
* ASA >Ⅲ.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative cognitive function | 1 month after the surgery.
  The incidence of POCD was compared between the experimental group and the control group.The preoperative and postoperative differences of the following scales were calculated and compared: Digit Span (forward and backward), Visual Retention and Paired Associate Verbal Learning subtests of the Wechsler Memory Scale, Digit Symbol subtest of the Wechsler Adult Intelligence ScaleRevised, Halstead-Reitan Trail Making Test (Part A), Corsi Block Test and Grooved Pegboard Test (favored and unfavored hand). The standard deviation (SD) for each test was computed from the preoperative scores. A participant whose postoperative performance declined by ≥1 SD as compared to each preoperative test score on ≥2 tests was classified as POCD.
Postoperative cognitive function | 3 months after the surgery.
  The incidence of POCD was compared between the experimental group and the control group.The preoperative and postoperative differences of the following scales were calculated and compared: Digit Span (forward and backward), Visual Retention and Paired Associate Verbal Learning subtests of the Wechsler Memory Scale, Digit Symbol subtest of the Wechsler Adult Intelligence ScaleRevised, Halstead-Reitan Trail Making Test (Part A), Corsi Block Test and Grooved Pegboard Test (favored and unfavored hand). The standard deviation (SD) for each test was computed from the preoperative scores. A participant whose postoperative performance declined by ≥1 SD as compared to each preoperative test score on ≥2 tests was classified as POCD.
Postoperative delirium | Consecutive 7 days after the surgery
  The incidence of POD was compared between the experimental group and the control group.Postoperative delirium was assessed by the Delirium Assessment Scale (CAM-ICU)
Acute postoperative pain | Consecutive 7 days after the surgery for acute pain
  The incidence of acute postoperative pain was compared between the experimental group and the control group.Acute postoperative pain was assessed by Visual Analogue Scale(VAS) for 7 consecutive days within 1 week after surgery.
Chronic Postsurgical pain | 3 months after the surgery for chronic pain
  The incidence of chronic postoperative pain (CPSP) was assessed by the Short Form McGill Pain Questionnaire (SF-MPQ) and Neuropathic Pain Scale (NPS).The incidence of CPSP was compared between the experimental group and the control group.

SECONDARY OUTCOMES:
TNF-α level in peripheral venous blood | 1 day before the surgery, Postoperative day 1, 3, 5
  The incidence of TNF-α level (pg/ml) in peripheral venous blood was compared between the experimental group and the control group
IL-6 level in peripheral venous blood | 1 day before the surgery, Postoperative day 1, 3, 5
  The incidence of IL-6 level (pg/ml) in peripheral venous blood was compared between the experimental group and the control group
IL-1β level in peripheral venous blood | 1 day before the surgery, Postoperative day 1, 3, 5
  The incidence of IL-1β level (pg/ml) in peripheral venous blood was compared between the experimental group and the control group
cortisol level in peripheral venous blood | 1 day before the surgery, Postoperative day 1, 3, 5
  The incidence of cortisol level (μg/dL) in peripheral venous blood was compared between the experimental group and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Yangzi Zhu, Doctor, Principal Investigator — Xuzhou Central Hospital; Liwei Wang, Doctor, Study Director — Xuzhou Central Hospital; Junli Cao, PhD & MD, Study Chair — Xuzhou Medical University; Daqing Ma, PhD & MD, Study Chair — Imperial College London
Locations (1):
- Xuzhou Central Hospital, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Glare P, Aubrey KR, Myles PS. Transition from acute to chronic pain after surgery. Lancet. 2019 Apr 13;393(10180):1537-1546. doi: 10.1016/S0140-6736(19)30352-6. PMID 30983589
- [Result] Lavand'homme P. Transition from acute to chronic pain after surgery. Pain. 2017 Apr;158 Suppl 1:S50-S54. doi: 10.1097/j.pain.0000000000000809. No abstract available. PMID 28134653
- [Result] Hovens IB, Schoemaker RG, van der Zee EA, Absalom AR, Heineman E, van Leeuwen BL. Postoperative cognitive dysfunction: Involvement of neuroinflammation and neuronal functioning. Brain Behav Immun. 2014 May;38:202-10. doi: 10.1016/j.bbi.2014.02.002. Epub 2014 Feb 8. PMID 24517920
- [Result] Eckenhoff RG, Maze M, Xie Z, Culley DJ, Goodlin SJ, Zuo Z, Wei H, Whittington RA, Terrando N, Orser BA, Eckenhoff MF. Perioperative Neurocognitive Disorder: State of the Preclinical Science. Anesthesiology. 2020 Jan;132(1):55-68. doi: 10.1097/ALN.0000000000002956. PMID 31834869
- [Result] Jin Z, Hu J, Ma D. Postoperative delirium: perioperative assessment, risk reduction, and management. Br J Anaesth. 2020 Oct;125(4):492-504. doi: 10.1016/j.bja.2020.06.063. Epub 2020 Aug 11. PMID 32798069
- [Result] Mohanty R, Lindroth H, Twadell S, Nair VA, Prabhakaran V, Sanders RD. A pilot study of neural correlates of perioperative executive function associated with noncardiac surgery in the elderly. Br J Anaesth. 2019 Nov;123(5):e517-e518. doi: 10.1016/j.bja.2019.08.001. Epub 2019 Aug 30. No abstract available. PMID 31474351
- [Result] Zhu Y, Zhou M, Jia X, Zhang W, Shi Y, Bai S, Rampes S, Vizcaychipi MP, Wu C, Wang K, Ma D, Yang Q, Wang L. Inflammation Disrupts the Brain Network of Executive Function after Cardiac Surgery. Ann Surg. 2023 Mar 1;277(3):e689-e698. doi: 10.1097/SLA.0000000000005041. Epub 2021 Jul 2. PMID 34225294
- [Result] Liu CH, Yang MH, Zhang GZ, Wang XX, Li B, Li M, Woelfer M, Walter M, Wang L. Neural networks and the anti-inflammatory effect of transcutaneous auricular vagus nerve stimulation in depression. J Neuroinflammation. 2020 Feb 12;17(1):54. doi: 10.1186/s12974-020-01732-5. PMID 32050990
- [Result] Huffman WJ, Subramaniyan S, Rodriguiz RM, Wetsel WC, Grill WM, Terrando N. Modulation of neuroinflammation and memory dysfunction using percutaneous vagus nerve stimulation in mice. Brain Stimul. 2019 Jan-Feb;12(1):19-29. doi: 10.1016/j.brs.2018.10.005. Epub 2018 Oct 9. PMID 30337243
- [Result] Redgrave J, Day D, Leung H, Laud PJ, Ali A, Lindert R, Majid A. Safety and tolerability of Transcutaneous Vagus Nerve stimulation in humans; a systematic review. Brain Stimul. 2018 Nov-Dec;11(6):1225-1238. doi: 10.1016/j.brs.2018.08.010. Epub 2018 Aug 23. PMID 30217648
- [Result] Farmer AD, Strzelczyk A, Finisguerra A, Gourine AV, Gharabaghi A, Hasan A, Burger AM, Jaramillo AM, Mertens A, Majid A, Verkuil B, Badran BW, Ventura-Bort C, Gaul C, Beste C, Warren CM, Quintana DS, Hammerer D, Freri E, Frangos E, Tobaldini E, Kaniusas E, Rosenow F, Capone F, Panetsos F, Ackland GL, Kaithwas G, O'Leary GH, Genheimer H, Jacobs HIL, Van Diest I, Schoenen J, Redgrave J, Fang J, Deuchars J, Szeles JC, Thayer JF, More K, Vonck K, Steenbergen L, Vianna LC, McTeague LM, Ludwig M, Veldhuizen MG, De Couck M, Casazza M, Keute M, Bikson M, Andreatta M, D'Agostini M, Weymar M, Betts M, Prigge M, Kaess M, Roden M, Thai M, Schuster NM, Montano N, Hansen N, Kroemer NB, Rong P, Fischer R, Howland RH, Sclocco R, Sellaro R, Garcia RG, Bauer S, Gancheva S, Stavrakis S, Kampusch S, Deuchars SA, Wehner S, Laborde S, Usichenko T, Polak T, Zaehle T, Borges U, Teckentrup V, Jandackova VK, Napadow V, Koenig J. International Consensus Based Review and Recommendations for Minimum Reporting Standards in Research on Transcutaneous Vagus Nerve Stimulation (Version 2020). Front Hum Neurosci. 2021 Mar 23;14:568051. doi: 10.3389/fnhum.2020.568051. eCollection 2020. PMID 33854421